CLINICAL TRIAL: NCT01473771
Title: Caring Letters for Military Suicide Prevention: A Randomized Controlled Trial
Brief Title: Caring Letters for Military Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Telehealth and Technology (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: W81XWH-11-2-0123; MOMRP (Other Grant/Funding Number: W81XWH-11-2-0123)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Suicide; Suicide, Attempted
Keywords: Suicide; Suicide, Attempted
MeSH Terms: conditions — Suicide; Suicide, Attempted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caring Letter Condition (CL) (Experimental): In the Caring Letters (CL) group, participants will be emailed "letters" for two years on a planned schedule. The emailed letters are simple expressions of care and include standard contact information for available health care services.
  Interventions: Behavioral: Caring Letter (email)
- Usual Care (UC) (No Intervention): The participants in the Usual Care (UC) group will not receive the emails.

INTERVENTIONS:
Behavioral: Caring Letter (email) — Participants will be emailed "letters" for two years. The first letter will be sent one week afer discharge from the inpatient psychiatric unit. There will be four subsequent email letters sent every month starting from the day of discharge, then another four every two months. The last four email letters will be sent every three months for the remainder of the two year period.
  Other Names: CLP
  Arms: Caring Letter Condition (CL)

SUMMARY:
The purpose of this multi-site randomized controlled trial is to determine if the Caring Letters intervention is effective in preventing suicide and suicidal behaviors among U.S. Service Members and Veterans. The primary aim of this project is determine whether caring communications following inpatient psychiatric treatment reduce suicide and self-inflicted injuries among U.S. military personnel and Veterans. The investigators will also explore treatment utilization by comparing the frequency of treatment visits after enrollment into the study. The following specific hypotheses will be tested:

Hypothesis 1: During a two year follow-up after the index hospital discharge, the frequency of suicide will be lower among participants in the Caring Letters group compared to those in the Usual Care group.

Hypothesis 2: The frequency of medically admitted self-inflicted injuries will also be lower in the Caring Letters group compared to the Usual Care group.

Hypothesis 3: The time to suicidal act, among those who do subsequently exhibit one, will be longer among participants in the Caring Letters group compared to the Usual Care group.

DETAILED DESCRIPTION:
This social/ behavioral study is a five year multi-site randomized controlled trial that will compare the Caring Letters intervention (with usual care) to usual care without the caring letters. Participants will be recruited from inpatient psychiatry units of collaborating military and Veterans Affairs (VA) sites and randomized to either a group that receives letters (Caring Letters group) or a group that does not receive letters (Usual Care group). The methodology of the intervention is updated with emails instead of postal letters. This study fills an important gap in the evidence base for the Caring Letter intervention through a methodologically rigorous research design.

ELIGIBILITY:
Inclusion Criteria:

* Current psychiatric inpatients
* Possess an active email account
* Informed consent
* Active duty military, Veteran, Retiree, National Guard or Reserves status

Exclusion Criteria:

* Not competent to consent
* Adverse behavioral problems
* The primary psychiatric nurse or attending psychiatrist considers that study to be clinically inappropriate
* Currently under arrest/incarceration
* Involuntary committed for psychiatric care status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1319 (Actual)
Dates: Start 2011-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Suicide Mortality Rates | Study Completion (2 years)
  Death Certificates as recorded in the Center for Disease Control (CDC's) National Death Index Plus(NDI-Plus) will be reviewed. The Social Security Administration Master Death File will also be used.

SECONDARY OUTCOMES:
Time to Suicidal Behavior | Study Completion (2 years)
  This is a survey that will assess participant suicidal behaviors and medical/psychiatric treatment utilization over the previous two years.

CONTACTS AND LOCATIONS:
Overall Officials: David D Luxton, PhD, Principal Investigator — National Center for Telehealth and Technology
Locations (6):
- United States (5):
  - Palo Alto VAHCS, Palo Alto, California
  - Naval Medical Center San Diego (NMCSD), San Diego, California
  - Tripler Army Medical Center (TAMC), Honolulu, Hawaii
  - VA Western New York, Buffalo VA Medical Center, Buffalo, New York
  - National Center for Telehealth and Technology, Tacoma, Washington
- Landstuhl Regional Medical Center, Landstuhl, Germany

REFERENCES:
- [Background] Reger, MA, Luxton DD, Skopp, NA, Lee, JA, Gahm, GA. Department of Defense Suicide Event Report (DoDSER): Calendar Year 2008 Annual Report: National Center for Telehealth and Technology, Defense Centers of Excellence for Psychological Health and TBI; 2009
- [Background] Luxton, DD, Skopp, NA, Kinn, JT, Bush, NE, Reger, MA, Gahm, GA. Department of Defense Suicide Event Report: Calendar Year 2009 Annual Report. Edited by Defense Centers of Excellence for Psychological Health & TBI (DCoE) National Center for Telehealth & Technology (T2); 2010.
- [Background] National Violent Death Reporting System: Centers for Disease Control and Prevention; 2009
- [Background] Joiner TE, Van Orden KA. The interpersonal-psychological theory of suicidal behavior indicates specific and crucial psychotherapeutic targets. International Journal of Cognitive Psychology 2008;1(1):80-89.
- [Background] Carter GL, Clover K, Whyte IM, Dawson AH, D'Este C. Postcards from the EDge project: randomised controlled trial of an intervention using postcards to reduce repetition of hospital treated deliberate self poisoning. BMJ. 2005 Oct 8;331(7520):805. doi: 10.1136/bmj.38579.455266.E0. Epub 2005 Sep 23. PMID 16183654
- [Background] Fleischmann A, Bertolote JM, Wasserman D, De Leo D, Bolhari J, Botega NJ, De Silva D, Phillips M, Vijayakumar L, Varnik A, Schlebusch L, Thanh HT. Effectiveness of brief intervention and contact for suicide attempters: a randomized controlled trial in five countries. Bull World Health Organ. 2008 Sep;86(9):703-9. doi: 10.2471/blt.07.046995. PMID 18797646
- [Background] De Leo D, Dello Buono M, Dwyer J. Suicide among the elderly: the long-term impact of a telephone support and assessment intervention in northern Italy. Br J Psychiatry. 2002 Sep;181:226-9. doi: 10.1192/bjp.181.3.226. PMID 12204927
- [Background] Cedereke M, Monti K, Ojehagen A. Telephone contact with patients in the year after a suicide attempt: does it affect treatment attendance and outcome? A randomised controlled study. Eur Psychiatry. 2002 Apr;17(2):82-91. doi: 10.1016/s0924-9338(02)00632-6. PMID 11973116
- [Background] Vaiva G, Vaiva G, Ducrocq F, Meyer P, Mathieu D, Philippe A, Libersa C, Goudemand M. Effect of telephone contact on further suicide attempts in patients discharged from an emergency department: randomised controlled study. BMJ. 2006 May 27;332(7552):1241-5. doi: 10.1136/bmj.332.7552.1241. PMID 16735333
- [Background] Gray GC, Chesbrough KB, Ryan MA, Amoroso P, Boyko EJ, Gackstetter GD, Hooper TI, Riddle JR; Millennium Cohort Study Group. The millennium Cohort Study: a 21-year prospective cohort study of 140,000 military personnel. Mil Med. 2002 Jun;167(6):483-8. PMID 12099084
- [Background] Linehan MM, Comtois K. (1996). Lifetime Parasuicide History. University of Washington, Seattle, WA. Unpublished work.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Rudd MD. The prevalence of suicidal ideation among college students. Suicide Life Threat Behav. 1989 Summer;19(2):173-83. doi: 10.1111/j.1943-278x.1989.tb01031.x. PMID 2749860
- [Background] Luxton DD, Rudd MD, Reger MA, Gahm GA. A psychometric study of the Suicide Ideation Scale. Arch Suicide Res. 2011;15(3):250-8. doi: 10.1080/13811118.2011.589720. PMID 21827314
- [Background] Van Orden KA, Witte TK, Gordon KH, Bender TW, Joiner TE Jr. Suicidal desire and the capability for suicide: tests of the interpersonal-psychological theory of suicidal behavior among adults. J Consult Clin Psychol. 2008 Feb;76(1):72-83. doi: 10.1037/0022-006X.76.1.72. PMID 18229985
- [Background] Joiner, TE. Why People Die by Suicide. Cambridge, MA: Harvard University Press; 2005.
- [Background] Luxton DD, Kinn JT, June JD, Pierre LW, Reger MA, Gahm GA. Caring Letters Project: a military suicide-prevention pilot program. Crisis. 2012 Jan 1;33(1):5-12. doi: 10.1027/0227-5910/a000093. PMID 21940244
- [Background] Luxton DD, June JD, Comtois KA. Can postdischarge follow-up contacts prevent suicide and suicidal behavior? A review of the evidence. Crisis. 2013 Jan 1;34(1):32-41. doi: 10.1027/0227-5910/a000158. PMID 22846445
- [Result] Motto JA. Suicide prevention for high-risk persons who refuse treatment. Suicide Life Threat Behav. 1976 Winter;6(4):223-30. PMID 1023455
- [Result] Mahon MJ, Tobin JP, Cusack DA, Kelleher C, Malone KM. Suicide among regular-duty military personnel: a retrospective case-control study of occupation-specific risk factors for workplace suicide. Am J Psychiatry. 2005 Sep;162(9):1688-96. doi: 10.1176/appi.ajp.162.9.1688. PMID 16135629
- [Result] Kang HK, Bullman TA. Is there an epidemic of suicides among current and former U.S. military personnel? Ann Epidemiol. 2009 Oct;19(10):757-60. doi: 10.1016/j.annepidem.2009.05.004. Epub 2009 Jul 22. No abstract available. PMID 19628411
- [Result] Chun S, Lee Y. The experience of posttraumatic growth for people with spinal cord injury. Qual Health Res. 2008 Jul;18(7):877-90. doi: 10.1177/1049732308318028. PMID 18552315
- [Result] Kaplan MS, Huguet N, McFarland BH, Newsom JT. Suicide among male veterans: a prospective population-based study. J Epidemiol Community Health. 2007 Jul;61(7):619-24. doi: 10.1136/jech.2006.054346. PMID 17568055
- [Result] Motto JA, Bostrom AG. A randomized controlled trial of postcrisis suicide prevention. Psychiatr Serv. 2001 Jun;52(6):828-33. doi: 10.1176/appi.ps.52.6.828. PMID 11376235
- [Result] Comtois KA, Linehan MM. Psychosocial treatments of suicidal behaviors: a practice-friendly review. J Clin Psychol. 2006 Feb;62(2):161-70. doi: 10.1002/jclp.20220. PMID 16342292
- [Result] Wright KM, Cabrera OA, Bliese PD, Adler AB, Hoge CW, & Castro CA. Stigma and barriers to care in soldiers postcombat. Psychological Services 2009; 6, 108-116.
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617